CLINICAL TRIAL: NCT02914626
Title: Intravitreal Ranibizumab (Lucentis®) for Neovascular Glaucoma- a Randomized Controlled Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LEANDRO CABRAL ZACHARIAS (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, LEANDRO CABRAL ZACHARIAS, Attending - Department of Ophthalmology- University of Sao Paulo, University of Sao Paulo General Hospital
Organization: University of Sao Paulo General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USaoPauloGH 294.326
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Glaucoma, Neovascular; Ranibizumab
Keywords: Glaucoma, Neovascular; Ranibizumab; Intraocular pressure; anti-VEGF; intravitreal injection
MeSH Terms: conditions — Glaucoma, Neovascular | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranibizumab (Experimental): Standard of care therapy plus intravitreal ranibizumab injections
  Interventions: Drug: Intravitreal ranibizumab
- Control (Sham Comparator): Standard of care therapy
  Interventions: Drug: Intravitreal ranibizumab

INTERVENTIONS:
Drug: Intravitreal ranibizumab — Intravitreal ranibizumab injection
  Other Names: Lucentis

SUMMARY:
Neovascular glaucoma is a potentially blinding condition characterized by the growth of newvessels at the anterior part of the eye. This growth is driven by the overexpression of a protein called Vascular Endothelial Growth Factor (VEGF). That happens in diseases such as diabetic retinopathy or venous retinal occlusion, and lead to a fast increase in intraocular pressure (IOP). Traditional treatment include laser photocoagulation of the retina in order to decrease VEGF formation. The investigators postulate that the use of anti-VEGF intravitreal injections may accelerate recovery and decrease the need of surgery in cases of neovascular glaucoma.

DETAILED DESCRIPTION:
This is a prospective, randomized controlled study that aims to evaluate the efficacy of ranibizumab (Lucentis®) as an adjunct in the treatment of patients with neovascular glaucoma.

28 patients with neovascular glaucoma (14 in the study group and 14 in the control standard of care group) will be recruited at a single center- University of Sao Paulo Medical School General Hospital. A complete ophthalmologic exam will be carried out, including the obtention of an informed consent for eligible patients willing to participate on the study.

Patients will be randomly assigned to either standard of care- retinal laser photocoagulation and clinical management of intraocular pressure with drops, or standard of care plus intravitreal ranibizumab injections. Two injections will be performed 30 days apart. The patients will be followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* IOP greater than 24 mmHg
* Iris or anterior chamber neovascularization
* At least 120 degrees of opened anterior chamber angle

Exclusion Criteria:

* Visual acuity worse than counting fingers in the fellow eye
* No light perception in the treated eye
* Any ocular infectious disease
* Use of systemic steroids
* Lack of media transparency precluding laser photocoagulation
* Thromboembolic disease
* Known hypersensitivity to ranibizumab
* Female participants at childbearing age not using oral contraceptives
* Use of intravitreal anti-VEGF over the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure | 6 months

SECONDARY OUTCOMES:
Anterior segment neovascularization | 6 months
Best corrected visual acuity | 6 months
Number of drugs needed for IOP control | 6 months
Need for IOP control surgery | 6 months

REFERENCES:
- [Derived] Rittiphairoj T, Roberti G, Michelessi M. Anti-vascular endothelial growth factor for neovascular glaucoma. Cochrane Database Syst Rev. 2023 Apr 3;4(4):CD007920. doi: 10.1002/14651858.CD007920.pub4. PMID 37010901